CLINICAL TRIAL: NCT04416659
Title: Flow Arrest Safety and Technical Success With Balloon Guide Catheters
Acronym: FAST-BGC
Status: Completed | Type: Observational
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Responsible Party: Sponsor
Other Study IDs: 3002
Record Dates: First submitted 2020-05-21; First posted 2020-06-04 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Neuro-vascular access — Adjunctive device providing a conduit for retrieval device during thrombectomy

SUMMARY:
The objective of this post-market registry is to assess technical efficacy and safety associated with the use of the BOSS Balloon Guide Catheter during neuro-vascular procedures while providing temporary arrest of blood flow.

DETAILED DESCRIPTION:
This is a prospective, multi-center, non-randomized observational registry evaluating use of BOSS balloon guide catheters in patients diagnosed with an acute ischemic stroke due to large intracranial vessel occlusion.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke vessel occlusion (ICA, M1 or M2) of the anterior circulation with associated symptoms
* Adult patient willing to provide Informed Consent
* Pre-treatment National Institutes of Health Stroke Scale (NIHSS) ≥ 6

Exclusion Criteria:

* Posterior circulation stroke
* Tandem occlusions
* Cervical carotid stenosis
* Participating in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Safety Evaluation | Hospital discharge or 7 days
  Incidence of device-related adverse events
Performance Evaluation | Completion of procedure
  Technical success of the BGC during procedure which includes inflation, deflation, retraction, flow arrest and reestablishment

CONTACTS AND LOCATIONS:
Overall Officials: Biraj Patel, MD, Principal Investigator — Carilion Clinic
Locations (9):
- United States (9):
  - BNI (St. Joseph's Hospital-Dignity Health), Phoenix, Arizona
  - Swedish-RIACO, Englewood, Colorado
  - Baptist Health Jacksonville, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - KUMC, Kansas City, Kansas
  - UMass Medical School, Worcester, Massachusetts
  - University of Missouri, Columbia, Missouri
  - Ft Sanders Regional Medical Center, Knoxville, Tennessee
  - Carilion Clinic, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No
No IPD will be available.